CLINICAL TRIAL: NCT07344727
Title: Impact of Haskap Berries on Recovery From High Intensity Resistance Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Collaborators: Montana State Agricultural Experiment Station (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2025-2138
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Inflammation; Oxidative Stress; Resistance Exercise; Recovery; Exercise Performance Recovery
Keywords: exercise performance; resistance exercise; recovery; oxidative stress; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Placebo and haskap interventions were designed to be comparable in taste, carbohydrate content, and appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Control (Placebo Comparator): The placebo supplement will have no polyphenol content and will be carbohydrate-matched to the experimental group. A twice daily dose (10-12 hours apart) will be consumed for 11 days.
  Interventions: Dietary Supplement: Placebo Comparator
- Haskap (Experimental): The haskap supplement will consist of a haskap berry smoothie. A twice daily dose (10-12) hours apart will be consumed for 11 days.
  Interventions: Dietary Supplement: Haskap berry smoothie

INTERVENTIONS:
Dietary Supplement: Haskap berry smoothie — A smoothie blend of berries and water
  Arms: Haskap
Dietary Supplement: Placebo Comparator — A smoothie with no polyphenolic content and matched in carbohydrate composition to the experimental haskap smoothie
  Arms: Placebo Control

SUMMARY:
The purpose of this clinical trial is to determine how certain food items affect oxidative stress, inflammation, and performance recovery from exercise induced muscle damage in a resistance trained population. The main questions The investigators aim to answer are the following:

* Do Haskaps speed the recovery of oxidative stress and inflammation markers after an intense lower body workout in resistance trained adults?
* Do Haskaps speed the recovery of performance measures after an intense lower body workout in resistance trained adults?
* The data collected in this investigation may also be used to ask additional questions not yet identified. For example, the investigators may use the stored samples to evaluate how the blood metabolites of participants differ before and after intense exercise. These additional questions are called secondary analyses. Please note that no genetic analysis will be conducted and racial and ethnic differences among participants will not be used in any secondary analyses.

Researches will compare Haskap juice to a color, flavor and carbohydrate matched placebo to see if Haskaps speed recovery in inflammation, oxidative stress and performance.

* Participants will be asked to drink either Haskap juice or placebo and follow a low polyphenolic diet
* Participants will perform an intense resistance workout
* Participants will have their blood drawn before and after the workout
* Performance will be analyzed at 24, 48 and 72 hours after the workout

DETAILED DESCRIPTION:
The main goal of the clinical trial is to learn more about how the haskap berry impacts the recovery process form intense resistance training. Haskap berries are very high in several compounds that function as antioxidants, such as polyphenols and vitamin C, which have many health promoting effects. For example, antioxidants lower inflammation and oxidative stress, which is known to cause damage to cells, proteins, and DNA. Oxidative stress is a result of excess free radicals, which are unstable molecules that can be created, along with inflammation, during intense exercise. This combination of excessive harmful byproducts in the body can cause soreness and decrease muscle performance experienced after a workout. However, the antioxidants in foods have the ability to neutralize free radicals that are produced and may reduce the time to recover from exercise.

To do this, a parallel, randomized, double blind, placebo controlled clinical trial of Haskap versus a placebo on resistance trained individuals will be completed. Participants will complete an intense workout consisting of barbell back squats and leg extension. Participants will drink either Haskap juice or placebo and follow a low polyphenolic diet for a total of 11 days. Participants will have their blood drawn before supplementation, before, immediately after and 8, 24, 48, and 72 hours after the workout to track recovery of blood markers. Performance will be analyzed via vertical jumps on force plates, maximal voluntary contraction of the quadriceps on a biodex, and speed of the squat at 24, 48, and 72 hours post workout.

ELIGIBILITY:
Inclusion Criteria:

* 2+ years of barbell squat experience
* Currently squatting at least once a week

Exclusion Criteria:

* BMI <18 or > 40 kg/m^2
* potential allergy to Haskap or placebo ingredients
* anti-inflammatory, weight loss, anabolic steroids, testosterone, or other drugs that may interfere with the measures of the study or any other medications that may interfere with study measures
* pregnant or lactating woman
* diagnosis with type 1 or type 2 diabetes, hypo-/hyperthyroidism or any other condition that may interfere with study measures
* smoke cigarettes
* lower extremity injury within the last year
* currently following a special diet including vegan, vegetarian, low carbohydrate, or ketogenic.
* currently consuming any of the following products: tart cherry juice, pomegranate juice, or 1 or more cups of acai or other berries per day.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Force Production | 72 hours
  Maximal Voluntary Contraction (MVC) to assess force production of knee extensors at 60 degrees.
Barbell Velocity | 72 hours
  Barbell velocity will be measure to determine how squat velocity recovers over the course of the study.
Vertical Jump | 72 hours
  Force plates will be used to evaluate vertical jump height.
Inflammation (pg/mL) | 11 days
  Serum interleukin (IL) IL-6, IL-10, IL-1ra, tumor necrosis factor alpha (TNF-alpha),
Lipid peroxidation | 11 days
  Plasma Malondialdehyde (MDA)
Creatine Kinase | 11 days
  Plasma
C-Reactive Protein | 11 days
  Plasma
Protein Carbonyls | 11 days
  Plasma

SECONDARY OUTCOMES:
Soreness | 72 hours
  Soreness will be evaluated objectively by participants drawing a line on a scale of 0-10 of how sore their legs are. 0 represents no soreness at all and 10 represents the most muscular soreness the participant has felt. A lower number could indicate less inflammation and muscular damage.
Acute Diet | 9 days
  24-hour dietary recall using the Automated Self-Administered 24-hour Dietary. Assessment Tool (ASA24). Outcome is macronutrient and micronutrient composition of food entry.
Sleep Questionnaire | 11 days
  Participants report information on the previous night's sleep. What time they went to sleep, how long it took them to fall asleep, how many hours they slept, whether these were normal sleep and wake times and how restful they perceive their sleep to be on a scale of 1 to 10. 1 indicates their sleep was not restful at all and 10 indicates their sleep was as restful as possible.

CONTACTS AND LOCATIONS:
Overall Officials: Mary P Miles, Principal Investigator — Montana State University
Locations (1):
- Montana State University, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-09-26): https://cdn.clinicaltrials.gov/large-docs/27/NCT07344727/Prot_ICF_000.pdf